CLINICAL TRIAL: NCT04047238
Title: Multicentre Randomized Controlled Study About the Effect of Individual Reminiscence Therapy on Cognition in Elderly People With Neurocognitive Disorder Attending Social Responses
Brief Title: Multicentre Study About the Effect of Individual Reminiscence Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rsocialform - Geriatria, Lda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01082019
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2019-08

CONDITIONS: Cognitive Impairment; Cognitive Decline; Dementia; Neurocognitive Disorders
Keywords: Dementia; Cognitive Impairment; Cognitive Decline; Neurocognitive Disorders; Elderly; Reminiscence Therapy; Individual Intervention; Cognition; Depression; Quality of Life
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Neurocognitive Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants who meet the inclusion criteria will be randomly assigned to the intervention group receiving Reminiscence Therapy or to a control group receiving treatment as usual. Participants in the intervention group will participate in two Reminiscence Therapy sessions per week for 3 months besides their treatment as usual. The sessions will be based on the Book of Past and Present and they will follow the same protocol in every participant institution.
  Interventions: Other: Reminiscence Therapy
- Control Group (No Intervention): Participants assigned to the control group will maintain their usual treatment in the institution, participating in the activities previously assigned to their individual care plan.

INTERVENTIONS:
Other: Reminiscence Therapy — Intervention group will receive two Reminiscence Therapy sessions per week for 3 months. Reminiscence therapy sessions will last approximately 50 minutes and will be developed according to the following structure:
  * Welcome to the patient and reality orientation therapy (7 minutes)
  * Conducting the main activity of reminiscence (40 minutes)
  * Closure, thank you for the participation and farewell until the next session (3 minutes) Reminiscence therapy sessions will have an individual format and will be conducted by a therapist previously trained in the protocol and the principles of Reminiscence Therapy. The Reminiscence activities of each session will be carried out following the protocol proposed in the Book of Past and Present.
  Arms: Intervention Group

SUMMARY:
This study aims to evaluate the effect of individual reminiscence therapy (RT) on the global cognitive function of people with neurocognitive disorders attending social responses and to evaluate the ability of individually applied reminiscence therapy (RT) to improve overall cognitive function, memory, executive function, mood and quality of life (QoL) of elderly people with neurocognitive impairment attending social responses. It is proposed a multicenter study with an experimental design with randomized controlled repeated measures. Participants in the intervention group will hold two RT sessions per week for three months. Control group participants will maintain their treatment as usual.

DETAILED DESCRIPTION:
Neurocognitive disorder is a major cause of disability among older people and its incidence is increasing due to an aging population. Neurocognitive disorders globally are estimated to affect 44.35 million people and it is expected that by the year 2050 the number of affected people globally will triple to 135.46 million.

The absence of effective pharmacological treatment that stops or slows down the development of the disease has aroused interest in non-pharmacological therapies as a complement to pharmacological treatment that may improve the quality of life of people with neurocognitive disorders. One of the most investigated and most traditional non-pharmacological therapy in this field is Reminiscence Therapy (RT).

RT involves discussing past activities, events and experiences, usually with the help of triggers, such as photographs, household objects and other familiar items from the past, music… that is, any object or stimulus that serves to stimulate remembrance. In its application to dementia, RT is based on the fact that the memory impairment of people with dementia means that they are able to recall events from their past life, especially from childhood to early adulthood, but cannot remember more recent facts. It focuses on preserved memories and abilities, promotes communication, and enables the person to connect with his/her past and regain his/her sense of personal identity. Thus, RT can be understood as an intervention on the edge of those of cognitive orientation and emotion-centered, with potential interactive effects on autobiographical memory and psychological well-being.

The investigators can distinguish at least two RT approaches. The first one is the "life review" where participants are guided through meaningful experiences from their biography trying to make sense of their life. This type of RT is more structured and is usually conducted in an individual format. It may imply the construction of "life books". This approach is considered to have an integrative function aimed at achieving a sense of validation, coherence and reconciliation with the person's past. Another approach is the simple reminiscence which involves the stimulation of autobiographical memory during conversations about specific themes of the past (such as holidays, food and drinks, work…) using stimuli that trigger memories. It has been described as an unstructured narrative of autobiographical memories. This reminiscence format can be conducted both individually and in groups and promotes communication between participants who share their memories and stories.

In any of the TR formats it is essential to introduce triggering stimuli (photographs, music, antique objects…) to aid in recall. These triggers may be generic, reflecting common experiences in the lives of people relevant to their age group (for example a textbook may serve to recall the experience during their school stage), or specific, with stimuli related to the individual's own experiences (for example photographs of an important life event such as your wedding day or a trip during your youth).

Regarding the effectiveness of RT, according to a recent Cochrane review, there is some evidence for its positive effects on cognition, QoL, communication, and possibly mood of people with dementia, although benefits are small. Despite the distinction between the two different approaches to RT (simple reminiscence vs. life review), the modality of therapy does not seem to be as important for positive effects as the individual or group format of the sessions and the context in which the intervention is administered (people who live in the community or people who are institutionalized).

According to the results of one review study, RT seems to be able to generate a small benefit on cognitive function immediately after the intervention, although it usually does not persist after a follow-up period. Regarding the administration format, individual RT effects seems slightly superior on cognition both immediately and after a follow-up period. In any case, its effects appear to be comparable to those of other cognitive stimulation therapies.

As for the effect of RT on QoL, a life-review-based individual RT study showed an improvement in Qol-AD. Effects with a group format do not seem consistent, showing little or no effect on QoL, although the key factor may be the application context (community vs. institution), with better results of group RT in institutionalized patients.

Group RT was associated with an effect on communication both after the intervention and at follow-up. This effect was not replicated in individual RT, with uncertain results.

Finally, despite evidence of the effect of RT on mood of older people without dementia, in the case of people with dementia only a small effect on mood was found for those participants. in individual RT.

Therefore, this research proposal aims to evaluate the ability of individual RT using a simple reminiscence format to improve the overall cognitive function, memory, executive function, mood and quality of life (QoL) of people with neurocognitive disorder attending social responses for the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnostic of a neurocognitive disorder according to the DSM-5 criteria.
* To have delivered the informed consent of the project, duly completed and signed, after prior information
* Capacity to communicate and understand.
* Possibility of gathering information about the participant's life history through their relatives or habitual caregivers, using the socio-familiar questionnaire design for that purpose.
* Being 65 years of age or older.
* Being a native Portuguese speaker.
* Regularly attend a social response institution that provides services for the elderly.

Exclusion Criteria:

* To suffer from an acute or severe illness that makes it impossible for them to participate in the intervention sessions.
* Serious sensory and physical limitations that prevent the participation in the sessions.
* Severe disconnection with the environment and very limited attention span.
* Presence of severe neuropsychiatric symptoms, such as hyperactivity, psychosis, severe depressive and anxiety symptoms and apathy, that prevent participation in the sessions or presence of uncontrolled delirium.
* Traumatic life history or marked by negative events relevant to the person that discourage the participation in the Reminiscence Therapy sessions.
* History of negative reactions during previous Reminiscence Therapy sessions or similar activities.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 251 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Cognitive functioning evaluated through Mini-Mental State Examination | Pre and post-intervention (3 months)
  Significant statistic improvement in the participant's test scores between pre-intervention assessment and post-intervention assessment. Mini-Mental State Examination is a brief cognitive screening test. Scores range between 0 - 30 points. Higher scores indicate better cognitive function.

SECONDARY OUTCOMES:
Memory funtion evaluated through Memory Alteration Test | Pre and post-intervention (3 months)
  Significant statistic improvement in the participant's test scores between pre-intervention assessment and post-intervention assessment. Memory Alteration Test is an easy and fast instrument that assesses five memory domains: orientation in time, short term memory, semantic memory, free recall and recall with clues. Scores range between 0 - 50 points. Higher scores indicate better memory.
Executive functions evaluated through Frontal Assessment Battery | Pre and post-intervention (3 months)
  Significant statistic improvement in the participant's test scores between pre-intervention assessment and post-intervention assessment. Frontal Assessment Battery assesses executive functions such as abstract thinking, mental flexibility, motor programming, interference sensibility, inhibitory control and environmental independence. Scores range between 0 - 18 points. Higher scores indicate better cognitive function.
Mood evaluated through Geriatric Depression Scale -15 | Pre and post-intervention (3 months)
  Significant statistic improvement in the participant's test scores between pre-intervention assessment and post-intervention assessment. Geriatric Depression Scale -15 is composed by 15 yes/no answer items and it has good psychometric characteristics to assess depression in older people. Scores range between 0 - 15 points. Higher scores indicate more severe depressive symptoms.
Quality of life evaluated through Quality of Life - Alzheimer's Disease | Pre and post-intervention (3 months)
  Significant statistic improvement in the participant's test scores between pre-intervention assessment and post-intervention assessment. Quality of Life - Alzheimer's Disease is an instrument to assess quality of life in people diagnosed with dementia, gathering information from the patient and the caregiver. It is composed by 13 items regarding perception of health, mood, functional abilities, interpersonal relationships and hobbies, decision making ability and life in general. It has good psychometric characteristics and it's use has been recommended to evaluate psychossocial interventions. Scores range between 13 - 52 points. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Susana I Justo Henriques, PhD, Principal Investigator — Cediara and University of de Santiago de Compostela; Enrique Pérez Sáez, PhD, Principal Investigator — CRE Alzheimer and University of Salamanca; João L Alves Apóstolo, PhD, Principal Investigator — Nursing School of Coimbra
Locations (25):
- Portugal (25):
  - Cediara - Assoc. Sol. Social de Ribeira de Fráguas, Albergaria-a-Velha, Aveiro District
  - Rsocialform - Geriatria, Lda., Mealhada, Aveiro District
  - Santa Casa Da Misericórdia de Ovar, Ovar, Aveiro District
  - Lar D. Pedro V, Praia da Vitória, Azores
  - Delicate Age Lda., Portimão, Faro District
  - APARSIN - Assoc. Port. de Apoio e Reabilitação Sénior de Intervenção Neurológica, Elvas, Portalegre District
  - Santa Casa Da Misericordia de Almada - Centro São Lázaro, Almada, Setúbal District
  - Centro Social Vale Do Homem, Braga
  - Santa Casa Da Misericórdia de Vila Verde, Braga
  - Centro Zulmira Pereira Simões, Braga
  - Santa Casa Da Misericórdia de Castelo Branco, Castelo Branco
  - Santa Casa Da Misericórdia de Vila Velha de Ródão, Castelo Branco
  - Centro Social Paroquial Dornelas, Guarda
  - Primavida Residência Sénior Amor, Leiria
  - Santa Casa Da Misericórdia de Alcobaça, Leiria
  - Santa Casa Da Misericórdia Do Alvorge, Leiria
  - Associação Alzheimer Portugal, Lisbon
  - Irmãs Hospitaleiras - Casa de Saúde Da Idanha, Lisbon
  - Centro Social de Tolosa, Portalegre
  - Centro Social Paroquial Recarei, Porto
  - Associação de Solidariedade Social S. Tiago de Rebordões, Porto
  - Santa Casa Da Misericordia de Coruche, Santarém
  - Santa Casa Da Misericórdia de Melgaço, Viana do Castelo
  - Santa Casa Da Misericórdia de Vouzela, Viseu
  - Pesqueiramiga- Associação de Solidariedade Social, Viseu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akanuma K, Meguro K, Meguro M, Sasaki E, Chiba K, Ishii H, Tanaka N. Improved social interaction and increased anterior cingulate metabolism after group reminiscence with reality orientation approach for vascular dementia. Psychiatry Res. 2011 Jun 30;192(3):183-7. doi: 10.1016/j.pscychresns.2010.11.012. Epub 2011 May 4. PMID 21543189
- [Background] Amieva H, Robert PH, Grandoulier AS, Meillon C, De Rotrou J, Andrieu S, Berr C, Desgranges B, Dubois B, Girtanner C, Joel ME, Lavallart B, Nourhashemi F, Pasquier F, Rainfray M, Touchon J, Chene G, Dartigues JF. Group and individual cognitive therapies in Alzheimer's disease: the ETNA3 randomized trial. Int Psychogeriatr. 2016 May;28(5):707-17. doi: 10.1017/S1041610215001830. Epub 2015 Nov 17. PMID 26572551
- [Background] Apóstolo JLA, Loureiro LMJ, Reis IAC, Silva IALL, Cardoso DFB, Sfetcu R. Contribution to the adaptation of the Geriatric Depression Scale -15 into Portuguese. Revista de Enfermagem Referência IV(3): 65-73, 2014. doi: 10.12707/RIV14033.
- [Background] Serrani Azcurra DJ. A reminiscence program intervention to improve the quality of life of long-term care residents with Alzheimer's disease: a randomized controlled trial. Braz J Psychiatry. 2012 Dec;34(4):422-33. doi: 10.1016/j.rbp.2012.05.008. PMID 23429813
- [Background] Barrios H, Verdelho A, Narciso S, Goncalves-Pereira M, Logsdon R, de Mendonca A. Quality of life in patients with cognitive impairment: validation of the Quality of Life-Alzheimer's Disease scale in Portugal. Int Psychogeriatr. 2013 Jul;25(7):1085-96. doi: 10.1017/S1041610213000379. Epub 2013 Mar 27. PMID 23534370
- [Background] Caddell LS, Clare L. The impact of dementia on self and identity: a systematic review. Clin Psychol Rev. 2010 Feb;30(1):113-26. doi: 10.1016/j.cpr.2009.10.003. PMID 19896760
- [Background] Charlesworth G, Burnell K, Crellin N, Hoare Z, Hoe J, Knapp M, Russell I, Wenborn J, Woods B, Orrell M. Peer support and reminiscence therapy for people with dementia and their family carers: a factorial pragmatic randomised trial. J Neurol Neurosurg Psychiatry. 2016 Nov;87(11):1218-1228. doi: 10.1136/jnnp-2016-313736. Epub 2016 Aug 12. PMID 27521377
- [Background] Dempsey L, Murphy K, Cooney A, Casey D, O'Shea E, Devane D, Jordan F, Hunter A. Reminiscence in dementia: a concept analysis. Dementia (London). 2014 Mar 1;13(2):176-92. doi: 10.1177/1471301212456277. Epub 2012 Aug 17. PMID 24599812
- [Background] Dubois B, Slachevsky A, Litvan I, Pillon B. The FAB: a Frontal Assessment Battery at bedside. Neurology. 2000 Dec 12;55(11):1621-6. doi: 10.1212/wnl.55.11.1621. PMID 11113214
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Gonzalez J, Mayordomo T, Torres M, Sales A, Melendez JC. Reminiscence and dementia: a therapeutic intervention. Int Psychogeriatr. 2015 Oct;27(10):1731-7. doi: 10.1017/S1041610215000344. Epub 2015 Mar 13. PMID 25765779
- [Background] Haight BK, Gibson F, Michel Y. The Northern Ireland life review/life storybook project for people with dementia. Alzheimers Dement. 2006 Jan;2(1):56-8. doi: 10.1016/j.jalz.2005.12.003. PMID 19595856
- [Background] Kirk M, Berntsen D. A short cut to the past: Cueing via concrete objects improves autobiographical memory retrieval in Alzheimer's disease patients. Neuropsychologia. 2018 Feb;110:113-122. doi: 10.1016/j.neuropsychologia.2017.06.034. Epub 2017 Jul 1. PMID 28676268
- [Background] Kirk M, Rasmussen KW, Overgaard SB, Berntsen D. Five weeks of immersive reminiscence therapy improves autobiographical memory in Alzheimer's disease. Memory. 2019 Apr;27(4):441-454. doi: 10.1080/09658211.2018.1515960. Epub 2018 Sep 8. PMID 30198380
- [Background] Lai CK, Chi I, Kayser-Jones J. A randomized controlled trial of a specific reminiscence approach to promote the well-being of nursing home residents with dementia. Int Psychogeriatr. 2004 Mar;16(1):33-49. doi: 10.1017/s1041610204000055. PMID 15190995
- [Background] Lima CF, Meireles LP, Fonseca R, Castro SL, Garrett C. The Frontal Assessment Battery (FAB) in Parkinson's disease and correlations with formal measures of executive functioning. J Neurol. 2008 Nov;255(11):1756-61. doi: 10.1007/s00415-008-0024-6. Epub 2008 Sep 25. PMID 18821046
- [Background] Moniz-Cook E, Vernooij-Dassen M, Woods R, Verhey F, Chattat R, De Vugt M, Mountain G, O'Connell M, Harrison J, Vasse E, Droes RM, Orrell M; INTERDEM group. A European consensus on outcome measures for psychosocial intervention research in dementia care. Aging Ment Health. 2008 Jan;12(1):14-29. doi: 10.1080/13607860801919850. PMID 18297476
- [Background] Morgado J, Rocha CS, Maruta C, Guerreiro M, Martins IP. Novos valores normativos do Mini-Mental State Examination. Sinapse 2: 10-16, 2009.
- [Background] O'Shea E, Devane D, Cooney A, Casey D, Jordan F, Hunter A, Murphy E, Newell J, Connolly S, Murphy K. The impact of reminiscence on the quality of life of residents with dementia in long-stay care. Int J Geriatr Psychiatry. 2014 Oct;29(10):1062-70. doi: 10.1002/gps.4099. Epub 2014 Mar 14. PMID 24633858
- [Background] Pinquart M, Duberstein PR, Lyness JM. Effects of psychotherapy and other behavioral interventions on clinically depressed older adults: a meta-analysis. Aging Ment Health. 2007 Nov;11(6):645-57. doi: 10.1080/13607860701529635. PMID 18074252
- [Background] Rami L, Molinuevo JL, Sanchez-Valle R, Bosch B, Villar A. Screening for amnestic mild cognitive impairment and early Alzheimer's disease with M@T (Memory Alteration Test) in the primary care population. Int J Geriatr Psychiatry. 2007 Apr;22(4):294-304. doi: 10.1002/gps.1672. PMID 16998781
- [Background] Sarkamo T, Tervaniemi M, Laitinen S, Numminen A, Kurki M, Johnson JK, Rantanen P. Cognitive, emotional, and social benefits of regular musical activities in early dementia: randomized controlled study. Gerontologist. 2014 Aug;54(4):634-50. doi: 10.1093/geront/gnt100. Epub 2013 Sep 5. PMID 24009169
- [Background] Subramaniam P, Woods B. Towards the therapeutic use of information and communication technology in reminiscence work for people with dementia: a systematic review. International Journal of Computers in Healthcare 1: 106-125, 2010. doi: 10.1504/IJCIH.2010.037457.
- [Background] Subramaniam P, Woods B. The impact of individual reminiscence therapy for people with dementia: systematic review. Expert Rev Neurother. 2012 May;12(5):545-55. doi: 10.1586/ern.12.35. PMID 22550983
- [Background] Subramaniam P, Woods B, Whitaker C. Life review and life story books for people with mild to moderate dementia: a randomised controlled trial. Aging Ment Health. 2014;18(3):363-75. doi: 10.1080/13607863.2013.837144. Epub 2013 Sep 24. PMID 24063317
- [Background] Tadaka E, Kanagawa K. Effects of reminiscence group in elderly people with Alzheimer disease and vascular dementia in a community setting. Geriatrics & Gerontology International 7: 167-173, 2007. doi: 10.1111/j.1447-0594.2007.00381.x.
- [Background] Thorgrimsen L, Schweitzer P, Orrell M. Evaluating reminiscence for people with dementia: A pilot study. The Arts in Psychotherapy 29: 93-97, 2002. doi: 10.1016/S0197-4556(01)00135-6.
- [Background] Westerhof GJ, Bohlmeijer E, Webster JD. Reminiscence and mental health: A review of recent progress in theory, research and interventions. Ageing & Society 30: 697-721, 2010. doi: 10.1017/S0144686X09990328.
- [Background] Wong PT, Watt LM. What types of reminiscence are associated with successful aging? Psychol Aging. 1991 Jun;6(2):272-9. doi: 10.1037//0882-7974.6.2.272. PMID 1863396
- [Background] Woods RT, Bruce E, Edwards RT, Hounsome B, Keady J, Moniz-Cook ED, Orrell M, Russell IT. Reminiscence groups for people with dementia and their family carers: pragmatic eight-centre randomised trial of joint reminiscence and maintenance versus usual treatment: a protocol. Trials. 2009 Jul 30;10:64. doi: 10.1186/1745-6215-10-64. PMID 19642992
- [Background] Woods RT, Bruce E, Edwards RT, Elvish R, Hoare Z, Hounsome B, Keady J, Moniz-Cook ED, Orgeta V, Orrell M, Rees J, Russell IT. REMCARE: reminiscence groups for people with dementia and their family caregivers - effectiveness and cost-effectiveness pragmatic multicentre randomised trial. Health Technol Assess. 2012;16(48):v-xv, 1-116. doi: 10.3310/hta16480. PMID 23211271
- [Background] Woods B, O'Philbin L, Farrell EM, Spector AE, Orrell M. Reminiscence therapy for dementia. Cochrane Database Syst Rev. 2018 Mar 1;3(3):CD001120. doi: 10.1002/14651858.CD001120.pub3. PMID 29493789
- [Background] Woods B, Spector A, Jones C, Orrell M, Davies S. Reminiscence therapy for dementia. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD001120. doi: 10.1002/14651858.CD001120.pub2. PMID 15846613
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Freitas S, Simoes MR, Alves L, Santana I. The Relevance of Sociodemographic and Health Variables on MMSE Normative Data. Appl Neuropsychol Adult. 2015;22(4):311-9. doi: 10.1080/23279095.2014.926455. Epub 2014 Dec 22. PMID 25531579
- [Background] Apóstolo JLA, Bobrowicz-Campos M, dos Reis IAC, Henriques SJ, Correia CAV. Exploring the screening capacity of the European Portuguese version of the 15-item Geriatric Depression Scale. Revista de Psicopatología y Psicología Clínica 23: 99-107, 2018. doi: 10.5944/rppc.vol.23.num.2.2018.21050.
- [Background] Guerreiro M, Silva AP, Botelho MA, Leitão O, Castro-Caldas A, Garcia. Adaptação à população portuguesa da tradução do Mini Mental State Examination (MMSE). Revista Portuguesa de Neurologia 1: 9-10, 1994.
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Quality of life in Alzheimer's disease: Patient and caregiver reports. Journal of Mental Health and Aging 5: 21-32, 1999.
- [Background] Morgan S, Woods RT. Life review with people with dementia in care homes: A preliminary randomized controlled trial. Non-pharmacological Therapies in Dementia 1: 43-60, 2010.